CLINICAL TRIAL: NCT06212141
Title: Clinical Comparison of Convetional Bulk-Fill Composite Resins and Thermoviscous Bulk-Fill Composite Resins in Class II Restorations
Brief Title: Comparison of Bulk-Fill Composite Resins in Class II Restorations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Meriç Tuncer, principle investigator, Hacettepe University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KA-22065
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Class II Dental Caries
Keywords: Bulk-Fill Composite; Thermoviscous Bulk-Fill Composite; Class II Restorations

STUDY DESIGN:
Intervention Model Description: Randomized split-mouth clinical trial
Who Masked: Outcomes Assessor
Masking Description: single-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VisCalor Bulk (Active Comparator): Thermoviscous Bulkfill composite resin Warming of the material makes it flowable for the application and then sculptable immediately afterwards (thermoviscous technology) Optimal flowing to margins and undercut regions One universal and three aesthetic shades Cannula form
  Interventions: Device: VisCalor Bulk,VOCO,Germany
- Admira Fusion x-tra (Active Comparator): Ormocer based bulkfill composite Purely ceramic-based, bulk fill restorative material Reliable curing of 4 mm layersby far the lowest polymerisation shrinkage (1.25 % by volume) and particularly low level of shrinkage stress, providing optimal marginal integrity.
  inert, so excellent biocompatible and extremely resistant to discolouration Easy handling, simple high-lustre polishing procedure coupled with high surface hardness guarantee first-class long-term results Universal shade with chameleon effect
  Interventions: Device: Admira Fusion x-tra,VOCO,Germany
- Filtek One Bulk (Active Comparator): Conventional bulkfill compositeFocused options powered by 3M technology help you complete posterior restorations in a single bulk placement.
  5 shades avaible : A1, A2, A3, B1, and C2. Excellent adaptation and sculptability for fast, easy placement. One-step placement : Tackle deep cavities with up to 5 mm depth of cure
  Interventions: Device: Filtek One Bulk,3M,Germany

INTERVENTIONS:
Device: VisCalor Bulk,VOCO,Germany — It was placed class II restorations.Before applying it, a 37% orthophosphoric acid will be injected into the cavity for 30 sec. on the enamel and 15 sec. on the dentin. Then, cavity will be rinsed with pressurized air and water for 15 sec. and Futura Bond U adhesive agent will be applied to the enamel and dentin surfaces using a disposable applicator for 20 sec. Then light air pressure will be applied for 5 sec., and then polymerization will be carried out for 10 sec. using LED light.
  When it comes to the application of VisCalor , the VisCalor Gun , heating device will be used. A disposable composite capsule will be placed into the device, and it will be heated by selecting program 1 (65°C) for 30 sec. The material will remain hot for 2.5 min.
  The nozzle of the capsule on the gun will be directly applied to the deepest part of the cavity, ensuring that the material is placed from bottom to top without exceeding 4 mm. Polymerization will be carried out with LED for 10 sec.
  Arms: VisCalor Bulk
Device: Admira Fusion x-tra,VOCO,Germany — Admira Fusion x-tra composite resin was placed class II restorations. Before applying it an orthophosphoric acid with a concentration of 37% will be injected into the cavity for 30 sec. on the enamel and 15 sec. on the dentin. Then, cavity will be rinsed with pressurized air and water for 20 sec. And Futura Bond U adhesive agent will be applied to the enamel and dentin surfaces using a disposable applicator for 20 sec. Following the manufacturer's recommendations, light air pressure will be applied for 5 sec, and then polymerization will be carried out for 10 sec. using LED light with a power of 1200 mW/cm².
  Afterwards bulk-fill composite will be placed in the cavity, ensuring that each layer does not exceed 4 mm, and appropriate occlusal shaping will be performed. Polymerization will be carried out with LED light for 20 seconds.
  Arms: Admira Fusion x-tra
Device: Filtek One Bulk,3M,Germany — Filtek One Bulk composite resin was placed class II restorations. Before applyingthe material, a 37% orthophosphoric acid will be injected into the cavity for 30 sec. on the enamel and 15 sec. on the dentin, followed by rinsing the cavity with pressurized air and water for 20 sec.Then , adhesive agent will be applied to the enamel and dentin surfaces using a disposable applicator for 20 sec. Following the manufacturer's recommendations, light air pressure will be applied for 5 sec, and then polymerization will be carried out for 10 sec using LED light .
  Afterwards, bulk-fill composite will be placed in the cavity, ensuring that each layer does not exceed 4 mm, and appropriate occlusal shaping will be performed. Polymerization will be carried out with LED light at a power of 1200 mW/cm² for 10 sec from all directions, following the manufacturer's recommendations.
  Arms: Filtek One Bulk

SUMMARY:
The goal of this clinical trial is to evaluate the clinical performance of Class II restorations of a thermoviscous nanohybrid materials , of a bulk-fill composite resin, and of conventional nanohyribrid bulk-fill composite resins .

Class II restorations will be performed in patients using three different restorative materials.And restorations will be evaluated using modified US Public Health Service criteria Resorations will be photograped and restorations will be evaluated for 6,12 months.

DETAILED DESCRIPTION:
The aim of this clinical study was to evaluate the clinical performance of Class II restorations of a thermoviscous nanohybrid materials , of a bulk-fill composite resin, and of conventional nanohyribrid bulk-fill composite resins.

Methods and Materials: Class II restorations will be performed in patients using three different restorative materials: VisCalor Thermoviscous Bulk-Fill (VCB; a thermoviscous nanohybrid bulk-fill composite resin) , Admira Fusion x-tra ( AFT: a conventional nanohybrid bulk-fill composite resin) and 3M Filtek One Bulk-Fill Restprative (FOB: a conventional bulk-fill nanocomposite ) Futura Bond U adhesive will be used for both conventional bulk-fill composite resin restorations and thermoviscous bulk-fill composite resin restorations.

Criteria for inclusion of patients in the study : Healthy individuals without any systemic disease, patients who is between 18 and 60 years old, patiens who brush their teeth 2 times a day,voluntary individuals who have agreed to participate in the study and signed the illuminated consent form, who have been given initial periodontal treatment.

Criteria for not inclusion of volunteers in research:Women who are pregnant or breastfeeding ,patienrs with advanced periodontial disease,patiens using a moving segmental prosthesis,patiens who have maloclusions,patiens who have bruxism,patients with known allergies to resin-based restorative materials and binding agents

The restorations will be evaluated using modified US Public Health Service criteria in terms of retention, color match, marginal discoloration, anatomic form, marginal adaptation, secondary caries, postoperative sensitivity, and surface texture. Resorations will be photograped and restorations will be evaluated for 6,12 months

.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals without any systemic disease
* Patients who is between 18 and 60 years old,
* Patiens who brush their teeth 2 times a day
* Voluntary individuals who have agreed to participate in the study and signed the illuminated consent form, who have been given initial periodontal treatment.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Patients with advanced periodontial disease
* Patiens using a moving segmental prosthesis
* Patiens who have maloclusions,
* Patiens who have bruxism,
* Patients with known allergies to resin-based restorative materials and binding agents

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Marginal Adaptation | From baseline to 18 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding marginal adaptation. Marginal adaptation was evaluated by an independent clinician. Visual inspection with a mirror was performed . Scores; Alfa: Closely adapted, no visible crevice. Bravo: Visible crevice, explorer will penetrate. Charlie: Crevice in which dentin is exposed
Marginal Staining | From baseline to 18 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding marginal staining. Marginal staining was evaluated by an independent clinician. Visual inspection with a mirror was performed . Scores: Alfa: No discoloration. Bravo: Discoloration without. Charlie: Discoloration with penetration in pulpal direction
Retention | From baseline to 18 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by an independent clinician. Scores: Alfa: No loss of restorative material. Charlie: Any loss of restorative material
Seconder caries | From baseline to 18 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by an independent clinician. Scores: Alfa: No caries present. Charlie: Caries present
Postoperative sensitivity | From baseline to 18 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by an independent clinician. Scores: Alfa: Not present. Bravo: sensitive but diminishing in intensity. . Charlie:constant sensitivity, not diminishing in intensity

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Meserret Başeren, Prof.Dr., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Chesterman J, Jowett A, Gallacher A, Nixon P. Bulk-fill resin-based composite restorative materials: a review. Br Dent J. 2017 Mar 10;222(5):337-344. doi: 10.1038/sj.bdj.2017.214. PMID 28281590